CLINICAL TRIAL: NCT03038516
Title: 'Palliative-D' Vitamin D Supplementation to Palliative Cancer Patients - A Double Blind, Randomised Controlled Trial
Brief Title: 'Palliative-D' Vitamin D to Palliative Cancer Patients
Acronym: Palliative-D
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Linda Björkhem-Bergman, MD, PhD, Assoc Prof, Senior Consultant, Region Stockholm
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Palliative-D
Record Dates: First submitted 2017-01-17; First posted 2017-01-31 (Estimated); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin D (Active Comparator): Cholecalciferol (Detremin) solved in MIGLYOL® 812
  Interventions: Drug: Cholecalciferol
- Placebo (Placebo Comparator): MIGLYOL® 812
  Interventions: Device: Placebo

INTERVENTIONS:
Drug: Cholecalciferol — To test the hypothesis that vitamin D treatment during 12 weeks to palliative cancer patients is superior to placebo in decreasing opioid consumption, fatigue and infectious burden and increase quality of life.
  Other Names: Detremin
  Arms: Vitamin D
Device: Placebo — To test the hypothesis that placebo is inferior to vitamin D treatment during 12 weeks to palliative cancer patients in decreasing opioid consumption,
  Other Names: MIGLYOL® 812
  Arms: Placebo

SUMMARY:
To test the hypothesis that vitamin D treatment during 12 weeks to palliative cancer patients can decrease opioid consumption, fatigue and infectious burden and increase quality of life.

DETAILED DESCRIPTION:
PROTOCOL IDENTITY AND OBJECTIVES: EudraCT Number 2017-000268-14 Protocol Title: Vitamin D supplementation to palliative cancer patients - A double blind, randomised controlled trial. Acronym: "Palliative-D" Trial Objectives: To test the hypothesis that vitamin D treatment during 12 weeks to palliative cancer patients can decrease opioid consumption, fatigue and infectious burden and increase quality of life.

INVESTIGATIONAL MEDICINAL PRODUCTS (IMP): Test ProductDetremin, MA holder Renapharma; Pharmaceutical Form: Oil Route of Administration: Oral route

METHODOLOGY Trial Design: Double-blind, parallel randomised and placebo controlled trial Dose/Duration 4000 IU/day for 12 weeks

Primary Endpoint:

The decline of opioid-consumption during 12 weeks in the vitamin D group compared to the placebo group, based on 3 measurements with 4 weeks intervals.

Secondary end Points:

1. Decline in antibiotic consumption
2. Improvement in quality of life
3. Improvement in fatigue
4. Vitamin D levels in serum after 12 weeks
5. Association between opioid dose and genetic polymorphism in genes involved in the effect and metabolism of vitamin D in the body.

Efficacy Parameters:

Opioid dose, translated to fentanyl per hour measured at baseline and at week 4,8 and 12.

Antibiotic consumption expressed as % of days with antibiotics during the last 4 weeks measured at baseline and at week 4, 8 and 12.

Quality of Life measured with EORTC-QLQ-C15-PAL at baseline and after 12 weeks. Fatigue measured with EORTC-QLQ-C15-PAL at baseline and after 12 weeks. 25-hydroxyvitamin D levels in blood at baseline and after 12 weeks. ESAS (Edmonton Symptom Assessment Scale ) measured at baseline and at week 4, 8 and 12.

Safety Parameters: S-calcium will be controlled in all subjects at baseline, at week 4, 8 and 12 and U-calcium in selected cases Power: The least clinically meaningful effect is estimated to be a 20% decline in opioid dose compared to the placebo. To obtain this result with 80% power the number of patients is estimated to be 127 in each arm i.e. 254 patients in total. This includes a drop-out of 25% per group.

Statistical Analyse plan: The primary endpoint will be analysed using linear regression, using bias corrected and accelerated bootstrap confidence intervals, while controlling for baseline measure of opioid dose (similar to ANCOVA). Adjustment for other background variables - such as vitamin D-level at baseline, gender and age - will be made in a secondary analysis to gain efficiency. The continuous secondary endpoints will be analysed using the same method as the primary endpoint .

POPULATION OF TRIAL SUBJECTS Number of Subjects: 254 (127 vitamin D and 127 placebo) Description of Trial Subjects: Palliative Cancer Patients (any cancer form) with a life expectancy of more than 3 months.

TRIAL TIMETABLE First Subject In Aug 2017 Last Subject In Sept 2019 (25 months to include participants) Last Subject Out Dec 2019 End of intervention Dec 2019 End of follow up Dec2019 End of Trial: Dec 2020

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted to ASIH Stockholm Södra or Stockholms Sjukhem.
2. Incurable cancer patients with any type of cancer. They could have ongoing oncological treatment but only with palliative intention. No patients with ongoing oncological treatment with curative intended treated will be included.
3. The life expectancy should be at least 3 months according to the clinical assessment of the study physician at the screening visit.
4. The patient should have no cognitive failure, being able to comprehend oral and written information about the study.
5. 25 OHD < 50 nmol/L.
6. Men and women aged ≥18
7. Signed 'informed consent'

Exclusion Criteria:

1. Ongoing vitamin D supplementation at the time for inclusion.
2. Serum level of 25-OH vitamin D3 >50 nmol/L
3. Known sarkoidosis
4. Treatment with tiazides or digoxin or digitoxin
5. Primary hyperparathyroidism
6. Hypercalcaemia (verified by a laboratory result younger than 2 month)
7. Plans to leave the Stockholm county within 12 weeks of inclusion
8. History of kidney stones
9. Taking part of another clinical study involving drugs
10. Hypersensitivity to cholecalciferol and/or any of the excipients
11. Other criteria that could jeopardize the study or its intention as judged by the investigator
12. Not being able to perform EORTC-QLQ-C15-PAL or ESAS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-06-09 (Actual); Study Completion 2020-06-09 (Actual)

PRIMARY OUTCOMES:
Change in opioid dose during 12 weeks | 12 weeks
  The change in decline of opioid-consumption during 12 weeks in the vitamin D group compared to the placebo group, based on 4 measurements with 4 weeks intervals.

SECONDARY OUTCOMES:
Change in Antibiotic Consumption during 12 weeks | 12weeks
  Change in Antibiotic consumption expressed as % of days with antibiotics during the last 4 weeks measured at baseline and at week 4, 8 and 12.
Change in Quality of life after 12 weeks | 12 weeks
  Change in Quality of Life measured with EORTC-QLQ-C15-PAL at baseline and after 12 weeks.
Change in Fatigue after12 weeks | 12 weeks
  Change in Fatigue measured with EORTC-QLQ-C15-PAL at baseline and after 12 weeks.
Change in 25-hydroxyvitamin D levels after 12 weeks | 12 weeks
  Change in 25-hydroxyvitamin D levels in blood at baseline and after 12 weeks.
Change in Symptom burden during 12 weeks | 12 weeks
  Change in Symptom burden measured with ESAS (Edmonton Symptom Assessment Scale) at baseline and at week 4, 8 and 12.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Björkhem-Bergman, Assoc Prof, Principal Investigator — Stockholm Läns Landsting
Locations (3):
- Sweden (3):
  - ASIH Stockholm Norr, Solna, Stockholm County
  - ASIH Stockholm Södra, Älvsjö
  - Stockholms Sjukhem ASIH, Stockholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goodrose-Flores C, Bonn SE, Klasson C, Frankling MH, Lagerros YT, Bjorkhem-Bergman L. Appetite and its association with mortality in patients with advanced cancer - a Post-hoc Analysis from the Palliative D-study. BMC Palliat Care. 2023 Oct 26;22(1):159. doi: 10.1186/s12904-023-01287-1. PMID 37880704
- [Derived] Klasson C, Helde-Frankling M, Sandberg C, Nordstrom M, Lundh-Hagelin C, Bjorkhem-Bergman L. Vitamin D and Fatigue in Palliative Cancer: A Cross-Sectional Study of Sex Difference in Baseline Data from the Palliative D Cohort. J Palliat Med. 2021 Mar;24(3):433-437. doi: 10.1089/jpm.2020.0283. Epub 2020 Sep 16. PMID 32936046